CLINICAL TRIAL: NCT03228849
Title: Conservative Management Equally Effective to New Suture Anchor Technique for Acute Mallet Finger Deformity: A Prospective Randomized Clinical Trial
Brief Title: Comparison of New Suture Anchor Technique for Bony Mallet Injury Versus Conservative Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Hayati Durmaz, Professor, MD, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014/288
Record Dates: First submitted 2017-07-18; First posted 2017-07-25 (Actual); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Finger Injuries; Finger Fracture; Finger Mallet
Keywords: Bony mallet injury; Anchor suture; Conservative treatment; DIP joint
MeSH Terms: conditions — Finger Injuries | interventions — Conservative Treatment

STUDY DESIGN:
Intervention Model Description: Patients were randomly assigned to surgical or conservative groups. After 6 weeks patients in both groups were started on the same rehabilitation protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conservative Treatment (Active Comparator): Patients were treated with 6 weeks with splinting and were then started on physical therapy for 2 weeks.
  Interventions: Procedure: Conservative Treatment
- Surgical Treatment (Active Comparator): Patients were treated with the new suture anchor technique and after 6 weeks were started on physical therapy for 2 weeks.
  Interventions: Procedure: Suture anchor technique

INTERVENTIONS:
Procedure: Suture anchor technique — Suture anchors were used to attach bony fragment. On week 6, patients were then started on physical therapy for 2 weeks.
  Arms: Surgical Treatment
Procedure: Conservative Treatment — The injured finger was immobilized in an aluminium splint for 6 weeks. Patients were then started on physical therapy for 2 weeks.
  Arms: Conservative Treatment

SUMMARY:
This study aims to compare conservative treatment versus a new suture anchor technique for bony mallet finger in 29 patients.

DETAILED DESCRIPTION:
This study aims to compare conservative treatment versus a new suture anchor technique for bony mallet finger in 29 patients who presented to investigators' clinic between 2013 and 2015. Patients were randomly assigned to conservative or surgical treatment groups. Patients in the conservative group were followed with immobilization with aluminum splint and physical therapy. Patients in the surgical group were treated with investigators' new surgical suture anchor technique and then received physical therapy. The patients were followed for 12 months. Primary study outcomes were extension deficit, days to return to work and DIP flexion.

ELIGIBILITY:
Inclusion Criteria:

* Wehbe Schneider type 1 - 2 and type A - B fractures
* ability to provide closed reduction
* patients' voluntariness

Exclusion Criteria:

* Wehbe Schneider type C and type 3 fractures

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2015-06-15 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Extension deficit | 12 months
  The inability to actively extend DIP joint to 0 degrees.
DIP flexion | 12 months
  The maximum angle of flexion at DIP joint
Days to return to work | Starting from the date of the start of treatment until patients returns to work, assessed up to 12 months
  Time to return to work

CONTACTS AND LOCATIONS:
Overall Officials: Sefa Giray Batıbay, MD, Principal Investigator — Istanbul University
Locations (1):
- Istanbul University Faculty of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No consent was obtained from the patients specifically to share their participant data.

REFERENCES:
- [Background] Angermann P, Lohmann M. [Hand and wrist injuries. A study of 50.272 injuries]. Ugeskr Laeger. 1995 Feb 6;157(6):734-7. Danish. PMID 7701632
- [Background] Salazar Botero S, Hidalgo Diaz JJ, Benaida A, Collon S, Facca S, Liverneaux PA. Review of Acute Traumatic Closed Mallet Finger Injuries in Adults. Arch Plast Surg. 2016 Mar;43(2):134-44. doi: 10.5999/aps.2016.43.2.134. Epub 2016 Mar 18. PMID 27019806
- [Background] Eddy M. Hands, fingers, thumbs - assessment and management of common hand injuries in general practice. Aust Fam Physician. 2012 Apr;41(4):202-9. PMID 22472680
- [Background] Alla SR, Deal ND, Dempsey IJ. Current concepts: mallet finger. Hand (N Y). 2014 Jun;9(2):138-44. doi: 10.1007/s11552-014-9609-y. PMID 24839413
- [Background] Moss JG, Steingold RF. The long term results of mallet finger injury. A retrospective study of one hundred cases. Hand. 1983 Jun;15(2):151-4. doi: 10.1016/s0072-968x(83)80006-0. PMID 6884844
- [Background] Handoll HH, Vaghela MV. Interventions for treating mallet finger injuries. Cochrane Database Syst Rev. 2004;(3):CD004574. doi: 10.1002/14651858.CD004574.pub2. PMID 15266538
- [Background] Hamas RS, Horrell ED, Pierret GP. Treatment of mallet finger due to intra-articular fracture of the distal phalanx. J Hand Surg Am. 1978 Jul;3(4):361-3. doi: 10.1016/s0363-5023(78)80038-0. PMID 681720
- [Background] Smit JM, Beets MR, Zeebregts CJ, Rood A, Welters CFM. Treatment options for mallet finger: a review. Plast Reconstr Surg. 2010 Nov;126(5):1624-1629. doi: 10.1097/PRS.0b013e3181ef8ec8. PMID 21042117
- [Background] Toker S, Turkmen F, Pekince O, Korucu I, Karalezli N. Extension Block Pinning Versus Hook Plate Fixation for Treatment of Mallet Fractures. J Hand Surg Am. 2015 Aug;40(8):1591-6. doi: 10.1016/j.jhsa.2015.04.027. Epub 2015 Jun 10. PMID 26070233
- [Background] Lubahn JD. Mallet finger fractures: a comparison of open and closed technique. J Hand Surg Am. 1989 Mar;14(2 Pt 2):394-6. doi: 10.1016/0363-5023(89)90121-4. No abstract available. PMID 2732433
- [Background] Auchincloss JM. Mallet-finger injuries: a prospective, controlled trial of internal and external splintage. Hand. 1982 Jun;14(2):168-73. doi: 10.1016/s0072-968x(82)80011-9. No abstract available. PMID 6749606
- [Background] Garberman SF, Diao E, Peimer CA. Mallet finger: results of early versus delayed closed treatment. J Hand Surg Am. 1994 Sep;19(5):850-2. doi: 10.1016/0363-5023(94)90200-3. PMID 7806817
- [Background] Jones NF, Peterson J. Epidemiologic study of the mallet finger deformity. J Hand Surg Am. 1988 May;13(3):334-8. doi: 10.1016/s0363-5023(88)80003-0. PMID 3379264
- [Background] Nakamura K, Nanjyo B. Reassessment of surgery for mallet finger. Plast Reconstr Surg. 1994 Jan;93(1):141-9; discussion 150-1. PMID 8278469
- [Background] Panchal-Kildare S, Malone K. Skeletal anatomy of the hand. Hand Clin. 2013 Nov;29(4):459-71. doi: 10.1016/j.hcl.2013.08.001. PMID 24209945
- [Background] Valdes K, Naughton N, Algar L. Conservative treatment of mallet finger: A systematic review. J Hand Ther. 2015 Jul-Sep;28(3):237-45; quiz 246. doi: 10.1016/j.jht.2015.03.001. Epub 2015 Mar 10. PMID 26003015
- [Background] Valdes K, Naughton N, Algar L. ICF components of outcome measures for mallet finger: A systematic review. J Hand Ther. 2016 Oct-Dec;29(4):388-395. doi: 10.1016/j.jht.2016.06.005. Epub 2016 Oct 22. PMID 27780628
- [Background] Mak L, Aitkens LD, Novak CB. Mallet finger injuries-A new method to maintain distal interphalangeal joint extension. J Hand Ther. 2016 Jul-Sep;29(3):352-5. doi: 10.1016/j.jht.2016.01.002. Epub 2016 Feb 9. PMID 27496991
- [Background] Maitra A, Dorani B. The conservative treatment of mallet finger with a simple splint: a case report. Arch Emerg Med. 1993 Sep;10(3):244-8. doi: 10.1136/emj.10.3.244. PMID 8216604
- [Background] Saito K, Kihara H. A randomized controlled trial of the effect of 2-step orthosis treatment for a mallet finger of tendinous origin. J Hand Ther. 2016 Oct-Dec;29(4):433-439. doi: 10.1016/j.jht.2016.07.005. Epub 2016 Oct 18. PMID 27769840
- [Background] Stern PJ, Kastrup JJ. Complications and prognosis of treatment of mallet finger. J Hand Surg Am. 1988 May;13(3):329-34. doi: 10.1016/s0363-5023(88)80002-9. PMID 3379263
- [Background] Ulusoy MG, Karalezli N, Kocer U, Uysal A, Karaaslan O, Kankaya Y, Aslan C. Pull-in suture technique for the treatment of mallet finger. Plast Reconstr Surg. 2006 Sep;118(3):696-702. doi: 10.1097/01.prs.0000232983.23840.f2. PMID 16932181
- [Background] Phadnis J, Yousaf S, Little N, Chidambaram R, Mok D. Open reduction internal fixation of the unstable mallet fracture. Tech Hand Up Extrem Surg. 2010 Sep;14(3):155-9. doi: 10.1097/BTH.0b013e3181d13800. PMID 20818217
- [Background] Kim JY, Lee SH. Factors Related to Distal Interphalangeal Joint Extension Loss After Extension Block Pinning of Mallet Finger Fractures. J Hand Surg Am. 2016 Mar;41(3):414-9. doi: 10.1016/j.jhsa.2015.11.026. Epub 2016 Jan 12. PMID 26794127
- [Background] Husain SN, Dietz JF, Kalainov DM, Lautenschlager EP. A biomechanical study of distal interphalangeal joint subluxation after mallet fracture injury. J Hand Surg Am. 2008 Jan;33(1):26-30. doi: 10.1016/j.jhsa.2007.09.006. PMID 18261661
- [Background] Schneider LH. A biomechanical study of distal interphalangeal joint subluxation after mallet fracture injury. J Hand Surg Am. 2008 Sep;33(7):1248-9; author reply 1249. doi: 10.1016/j.jhsa.2008.04.014. No abstract available. PMID 18762129
- [Background] Crawford GP. The molded polythene splint for mallet finger deformities. J Hand Surg Am. 1984 Mar;9(2):231-7. doi: 10.1016/s0363-5023(84)80148-3. PMID 6715831
- [Background] Abouna JM, Brown H. The treatment of mallet finger. The results in a series of 148 consecutive cases and a review of the literature. Br J Surg. 1968 Sep;55(9):653-67. doi: 10.1002/bjs.1800550905. No abstract available. PMID 4877731
- [Background] Roh YH, Lee BK, Park MH, Noh JH, Gong HS, Baek GH. Effects of health literacy on treatment outcome and satisfaction in patients with mallet finger injury. J Hand Ther. 2016 Oct-Dec;29(4):459-464. doi: 10.1016/j.jht.2016.06.004. Epub 2016 Oct 17. PMID 27765527

DOCUMENTS (3):
  • Study Protocol (2013-05-23): https://cdn.clinicaltrials.gov/large-docs/49/NCT03228849/Prot_000.pdf
  • Informed Consent Form (2013-05-23): https://cdn.clinicaltrials.gov/large-docs/49/NCT03228849/ICF_001.pdf
  • Statistical Analysis Plan (2013-05-23): https://cdn.clinicaltrials.gov/large-docs/49/NCT03228849/SAP_002.pdf